CLINICAL TRIAL: NCT00997685
Title: A Single Arm, Open-label Phase II Study to Evaluate the Efficacy and Safety of Capecitabine Plus Oxaliplatin (XELOX) in the Peri-operative Treatment of Patients With Potentially Resectable Liver Metastasis From Colorectal Cancer
Brief Title: Evaluate Efficacy and Safety of XELOX in Potentially Resectable Liver Metastasis From Colorectal Cancer(CRC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Institutions of national drug clinical trials, Guangdong General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22298
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Potentially Resectable Liver Metastasis From CRC; Colorectal Cancer
Keywords: XELOX; potentially resectable liver metastasis from CRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine plus oxaliplatin，mCRC (Experimental)
  Interventions: Drug: Capecitabine plus oxaliplatin

INTERVENTIONS:
Drug: Capecitabine plus oxaliplatin — Xeloda: 1000mg/m2 bid, d1-14, q3w, Oxaliplatin:130mg/m2 d1, q3w,
  4 pre-operative cycles, 4 post-operative cycles
  Other Names: XELOX

SUMMARY:
This is a single arm, open-label phase II study to evaluate the efficacy and safety of Capecitabine plus oxaliplatin (XELOX) in the peri-operative treatment of patients with potentially resectable liver metastasis from colorectal cancer.

DETAILED DESCRIPTION:
To investigate the progression free survival (PFS) advantage of Xeloda plus oxaliplatin in the peri-operative treatment of potential resectable metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 and 65
* Histologically confirmed colorectal cancer and two methords of imaging detection confirmed liver metastasis
* Potentially curable by resection, as determined by a surgeon with hepatic surgery expertise
* No evidence of extrahepatic disease by chest x-ray or CT scan of the chest, abdomen, and pelvis
* Patients with adequate hepative, renal and bone marrow function
* Signed written informed consent

Exclusion Criteria:

* Pregnant or nursing patients (fertile patients must use effective contraception)
* Other malignancy within the past 5 years except completely resected nonmelanoma skin cancer or carcinoma in situ of the cervix
* Preexisting grade 2 or greater peripheral neuropathy
* Concurrent uncontrolled illness
* Ongoing or active infection
* Psychiatric illness or social situation that would preclude study compliance
* Less than 6 months since prior adjuvant fluorouracil-based chemotherapy
* Prior chemotherapy for liver metastasis
* Prior oxaliplatin for colorectal cancer
* Prior or concurrent hepatic artery infusion chemotherapy for metastatic disease
* Prior or concurrent radiotherapy for metastatic disease
* Prior or concurrent radiofrequency ablation for metastatic disease
* concurrent treatment with any other anti-cancer therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2009-11; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
To investigate the progression free survival (PFS) advantage of Xeloda plus oxaliplatin in the peri-operative treatment of potential resectable metastatic colorectal cancer | 3.6 years

SECONDARY OUTCOMES:
To investigate the response rate | 3.6 years
To evaluate the R0 resection rate | 3.6 years
To evaluate the safety profile of XELOX peri-operative treatment | 3.6 years

CONTACTS AND LOCATIONS:
Overall Officials: Feng Lin, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China